CLINICAL TRIAL: NCT05439239
Title: Effects of Hypoxic Repeated Sprint Training on Performance in Normoxia in Male and Female Athletes Participating in Team/Racket Sports
Brief Title: Effects of Hypoxic Repeated Sprint Training on Performance in Normoxia in Male and Female Athletes
Acronym: RSHwomen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RSH women
Record Dates: First submitted 2022-05-31; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Hypoxia; Repeated Sprints
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Single blind, parallel, gender-comparative, randomized controlled study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normoxic group females (Placebo Comparator): The participants in this group (12 females) will perform a repeated sprint training in normoxia.
  Interventions: Other: Repeated sprint training
- Hypoxic group females (Experimental): The participants in this group (12 females) will perform a repeated sprint training in hypoxia.
  Interventions: Other: Repeated sprint training
- Normoxic group males (Placebo Comparator): The participants in this group (12 males) will perform a repeated sprint training in normoxia.
  Interventions: Other: Repeated sprint training
- Hypoxic group males (Placebo Comparator): The participants in this group (12 males) will perform a repeated sprint training in hypoxia.
  Interventions: Other: Repeated sprint training

INTERVENTIONS:
Other: Repeated sprint training — Participants will perform 7 weeks of cycling repeated sprint training (2x/week). Inspired oxygen fraction (FiO2) will be set to 14.6% and 20.9% for the hypoxic and normoxic group to simulate an altitude of 3000 m and 300 m, respectively.
  The training sessions will consist of a 10-min warm up followed by 3 sets of 5 x 10-s all-out repeated sprints on the cycle ergometer. The number of sets will decrease to two during week 7. Participants will be instructed to try to reach and maintain maximal power output during each sprint. An active recovery at 30% of VO2max will be allowed for 20 s between sprints and for 5 min between sets. The training will end with a 10-min cool down at 30% VO2max. An individual fixed torque of 0.7 will be used during the sprints and it will be reduced to 0.5 Nm/kg at week 7.

SUMMARY:
With the increased participation of women in sports, it is essential to develop gender-tailored training strategies for improving exercise performance. Males and females exhibit gender-specific characteristics and they therefore respond differently to physical exercise. Improving repeated sprint ability (RSA, i.e., ability to perform repeated short duration sprints separated by brief recovery intervals) in women is important for sports performance, as it is a key factor in most team and racket sports. Repeated sprint training in hypoxia is increasingly popular in this field, as it has demonstrated further improvements in sea-level repeated sprint performance than similar training in normoxia. However, these observations are based mainly on male athletes. Whether the effects of hypoxic repeated sprint training on repeated sprint performance in normoxia differ between genders is not yet known, therefore the investigators propose to examine those possible differences in this study.

The aim of this study is to investigate whether the effects of hypoxic repeated sprint training on repeated sprint performance in normoxia differ between males and females who participate in team/racket sports.

Considering the sex-specific characteristics that males and females exhibit, the investigators hypothesize that after 7 weeks of hypoxic repeated sprint training the improvements in repeated sprint ability at sea level will be greater in males than in females.

To answer this question, the investigators will measure the following: body composition (lean body mass); body weight and height; VO2max; blood (estrogen, lactate, hemoglobin, hematocrit); repeated sprint ability (RSA) test; muscle oxygenation (concentrations for oxyhemoglobin, deoxyhemoglobin, and total hemoglobin/myoglobin); 30-s Wingate test; heart rate (HR); power output; rate of perceived exertion (RPE); visual analogue scale (VAS; pain level in legs).

The investigators will recruit 48 volunteers and they will randomly assign them into the normoxic or hypoxic training group, without giving any information about their group. The volunteers should meet the following inclusion criteria: females (on monophasic oral contraceptive pill) and males, age between 18-40 years, recreationally participating in team/racket sports min 3h/week with at least 2 years of experience prior to the study. Exclusion criteria will be: smoking, exposure to altitude >1500 m one month before the study, any health conditions or injuries that could compromise the participant's safety during training/testing, prescribed medication, performing repeated sprint training more than once per week.

Males and females, matched for VO2max and sprint performance, will perform repeated sprint training (3 sets during week 1-6, 2 sets during week 7 with 5min active recovery in between, 5 x 10s maximal sprints with 20s active recovery in between) in hypoxia or normoxia 2x/week for 7 weeks. Before and after the training period, the following tests and measurements will be performed: body composition analysis, VO2max test, blood sampling for measuring hemoglobin and estrogen concentrations and hematocrit, determination of hemoglobin mass, RSA test, muscle oxygenation assessment during RSA test, 30-s Wingate test and blood lactate measurements.

DETAILED DESCRIPTION:
A single blind, parallel, gender comparative, randomized controlled trial design will be used and the methodology of this study will be based on a previously applied successful protocol on males. Participants (males and females) will be randomly assigned to either the control group (repeated sprint training in normoxia; RSN) or the intervention group (repeated sprint training group in hypoxia; RSH), resulting in four groups in total (females RSN and RSH; males RSN and RSH). Due to the big number of participants required, the experiment will be split into two studies: RSN will be performed in study 1 and RSH in study 2. The experiment involves 7 weeks (week 1-7) of cycling repeated sprint training in normoxia or hypoxia, 2x/week, and two testing sessions before (week -2/-1, Pre-testing) and after (week 8/9, Post-testing) the training period. During the testing sessions, participants will complete the following exercise performance tests and measurements in normoxia: body composition assessment through DEXA (dual energy x-ray absorptiometry) and skinfold measurements, VO2max test, blood sampling at rest to measure hemoglobin and estrogen concentrations and hematocrit, determination of hemoglobin mass, repeated sprint ability (RSA) test and near-infrared spectroscopy (NIRS) measurement for muscle oxygenation, and 30-s Wingate test. Blood lactate will be measured at rest before and immediately after the following exercise performance tests: RSA and Wingate.

Preliminary visit:

During the week before Pre-testing, participants will be assessed for eligibility through a medical screening and completion of questionnaires (medical screening and physical activity/lifestyle questionnaires), after signing the informed consent related to the Pre-screening. If they are eligible and still wish to take part to the study, participants will sign the informed consent related to the study and they will get familiarized with all the experimental procedures.

Supervised training:

Participants will perform 7 weeks of cycling repeated sprint training (2x/week), starting the week after the Pre- testing and finishing the week before the Post-testing. The training sessions will take place in a hypoxic chamber consisting of a compressor, built in the laboratory. Inspired oxygen fraction (FiO2) will be set to 14.6% and 20.9% for RSH and RSN to simulate an altitude of 3000 m and 300 m, respectively. In order to blind subjects to altitude, the compressor system will also be running for RSN but with a normoxic airflow into the chamber. Temperature in the chamber will be maintained constant throughout the training program.

The training sessions will consist of a 10-min warm up at 50% of the VO2max of each participant, followed by 3 sets of 5 x 10-s all-out repeated sprints on the cycle ergometer. The number of sets will decrease to two during week 7. Participants will be instructed to try to reach and maintain maximal power output during each sprint. An active recovery at 30% of VO2max will be allowed for 20 s between sprints and for 5 min between sets. The training will end with a 10-min cool down at 30% VO2max. An individual fixed torque of 0.7 Nm/kg will be used during the sprints and it will be reduced to 0.5 Nm/kg at week 7. Power output and heart rate will be recorded during each training session. Water will be provided to all participants to ensure appropriate hydration during training. After each session, participants will be asked to report their rate of perceived exertion (RPE, Borg Scale, 6-20) and the level of pain in the legs (continuous visual analogic scale, VAS). At least one day of rest will be allowed between the two weekly sessions, to ensure optimal recovery. Participants will be asked to maintain their usual training outside the laboratory and fill a training diary.

Pre- and Post- testing:

Each pre- and post- testing session consists of two days. Participants will be asked to complete a food diary during the three days prior to each test session and reproduce their diet as much as possible. They will also be instructed to refrain from alcohol and caffeine intake during the 24 h before each test, and from heavy exercise during the 48 h before. Participants will be advised to consume a standard meal before the tests. During the tests, tap water will be provided ad libitum to all participants.

During testing day 1, body weight and height will be measured, and body composition will be assessed using DEXA (dual energy x-ray absorptiometry) scan and skinfold measurements. A blood sample will be taken at rest from the antecubital vein for measuring hemoglobin and estrogen concentrations, and hematocrit. Estrogen levels will also be assessed, to ensure that female participants are not ovulating (despite the pill) on the test days. Participants will then perform a maximal incremental exercise test to assess aerobic performance (VO2max). One hour after the test, hemoglobin mass will be determined according to the CO rebreathing method.

During testing day 2, participants will perform an RSA test and a Wingate test. Blood lactate concentration will be measured from an earlobe sample of 5ul at rest before each test and then immediately after and at 2, 4 and 6 minutes after the exercise performance tests, i.e., RSA and Wingate tests.

For all performance tests the participants will use the cycle ergometer. The seat and handlebar positions will be adjusted for each participant and reproduced for all tests. During the RSA and Wingate tests the investigators will record heart rate, peak and average power output, and pedaling frequency. After each test, participants will be asked to report their RPE and VAS.

Pre- and Post- testing will be performed in the exact same order in normoxia in the well-ventilated laboratory at a constant temperature of ~ 18 o C.

VO2max test

After blood sampling on day 1, participants will perform a VO2max test. The starting load for the test will be set at 1.2 W/kg LBM and will be incremented by 0.6 W/kg LBM every 2 min until exhaustion. Oxygen consumption and carbon dioxide production will be measured throughout the test using a gas exchange analyser, and maximum oxygen consumption (VO2max) will be determined. Heart rate will also be recorded during the test. Upon completion of the test, participants will be asked to report their RPE and VAS.

Repeated Sprint Ability Test

During testing day 2, participants will arrive at the laboratory and a baseline measurement (3min) of muscle oxygenation of the right vastus lateralis will be taken in a seated position using the NIRS method. Then participants will perform a 10-min warm-up at 50% of their VO2max, including two 5-s all-out sprints against a fixed torque of 0.8 Nm/kg. Following the warm-up, another NIRS measurement will be taken at rest. Participants will then start pedaling for 20 s at 30% VO2max before performing the RSA test. The test consists of 10-s all-out sprints against a fixed torque of 0.8 Nm/kg with a 20-s active recovery after each sprint at 30% VO2max. Participants will be instructed to try to reach and maintain maximal power output during each sprint of the test. They will also be given strong verbal encouragement and will be instructed to perform as many sprints as possible until volitional exhaustion. No indication on the number of sprints performed will be given. A minimal pedaling frequency of 70 rpm for more than 5 s during a sprint will be a criterion to stop the test. Upon completion of the test, a 10-min cool down at 30% VO2max will follow.

NIRS

Changes in muscle oxygenation will be measured during the RSA test by the NIRS technique using the difference in absorption characteristics of light between 760 and 850 nm. Skinfold will be measured with a caliper in order to confirm that the distance between the NIRS apparatus and the muscle is not higher than 16 mm. The apparatus will then be fixed on vastus lateralis of the right leg with a large bandage to avoid interference by extraneous light and loss of transmitted light out of the field of investigation.

Concentrations for oxyhemoglobin ([O2Hb]), deoxyhemoglobin ([HHb]) and total hemoglobin/myoglobin ([tHb]) will be determined. Amplitudes during the following sprints and the average value for all sprints throughout the RSA test (i.e. Δ[HHb]av and Δ[tHb]av) will be calculated. The same analysis will be performed during the successive recovery phases. In addition, the Δ[tHb]/Power will be calculated as the ratio between Δ[tHb] and mean power for each sprint as an index of blood perfusion relative to the intensity of each sprint.

Hemoglobin mass measurement

For this measurement, 7 blood samples of about 70ul will be taken at the fingertip, 5 before CO inhalation and 2 after. The CO-rebreathing method consists in the inhalation of a low quantity of CO (1m/kg bw) mixed with oxygen. Having a high affinity for hemoglobin, CO binds to the later preferentially. To measure total hemoglobin mass, the fraction of CO bound to hemoglobin (ABL90 Flex, Radiometer) will be evaluated before and after the inhalation of the mixed gas (oxygen + CO) as well as the CO concentration in the exhaled air (CO-meter, Dräger).

30 s Wingate Test

One hour after the RSA test, participants will perform a 10-min warm-up on the cycle ergometer at 30% of their VO2max including two 5-s sprints at a test load. Then they will complete a 30-s maximal cycling exercise with a resistance set to 7.5% of the participant's body weight (0.075 kg/kg bw). The participants will be asked to try and generate the highest power possible throughout the test and will receive strong verbal encouragement. A 10-min cool down will follow.

The investigators will match the male and female participants as closely as possible for sprint performance recorded during the RSA test of Pre- testing. The average power of the best two sprints will be calculated in Watts and then expressed as joules per kilogram of lean body mass (LBM). Moreover, the investigators will match participants for VO2max relative to LBM, recorded during the incremental test of Pre- testing.

ELIGIBILITY:
Inclusion Criteria:

* Females (on monophasic oral contraceptive pill)
* Males
* Must recreationally participating in team/racket sports min 3h/week with at least 2 years of experience prior to the study

Exclusion Criteria:

* Smoking
* Exposure to altitude >1500 m one month before the study
* Any health conditions or injuries that could compromise the participant's safety during training/testing
* Prescribed medication
* Performing repeated sprint training more than once per week.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Repeated sprint cycling performance in normoxia in males and females who participate in team or racket sports. | The primary outcome will be assessed twice for each participant: one time before the training program and one time after the training program. Testing will last no more than one hour.
  Performance will be determined through a repeated sprint ability test on the cycle ergometer, by the number of sprints and the power output during the sprints.
  The repeated sprint cycling performance will be assessed before and after a 7-week training program of repeated sprints in normoxia or hypoxia.

SECONDARY OUTCOMES:
Endurance capacity assessed using a maximal effort test on the cycle ergometer, namely VO2max test. | The secondary outcomes will be assessed twice for each participant: one time before the training program and one time after the training program.
  Endurance capacity will be measured in ml/min/lean body mass.
Lean body mass assessed by the DEXA scan. | The secondary outcomes will be assessed twice for each participant: one time before the training program and one time after the training program
  Expressed in kilos.
Fat percentage measured using the skinfolds method and the DEXA scan. | The secondary outcomes will be assessed twice for each participant: one time before the training program and one time after the training program
  Expressed as a percentage.
Hemoglobin mass measured using the CO rebreathing method. | The secondary outcomes will be assessed twice for each participant: one time before the training program and one time after the training program
  Hb mass will be expressed in g/kg.
Hemoglobin concentration measured using the HORIBA hematology analyzer. | The secondary outcomes will be assessed twice for each participant: one time before the training program and one time after the training program
  Expressed in g/dL.
Hematocrit measured using the HORIBA hematology analyzer. | The secondary outcomes will be assessed twice for each participant: one time before the training program and one time after the training program
  Expressed as a percentage.
Anaerobic capacity measured by the 30 s Wingate test on the cycle ergometer. | The secondary outcomes will be assessed twice for each participant: one time before the training program and one time after the training program
  Anaerobic capacity will be determined by the power output recorded during the test.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Physiology Lab, Louvain-la-Neuve, Brabant Walloon, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faiss R, Leger B, Vesin JM, Fournier PE, Eggel Y, Deriaz O, Millet GP. Significant molecular and systemic adaptations after repeated sprint training in hypoxia. PLoS One. 2013;8(2):e56522. doi: 10.1371/journal.pone.0056522. Epub 2013 Feb 20. PMID 23437154
- [Background] Costello JT, Bieuzen F, Bleakley CM. Where are all the female participants in Sports and Exercise Medicine research? Eur J Sport Sci. 2014;14(8):847-51. doi: 10.1080/17461391.2014.911354. Epub 2014 Apr 25. PMID 24766579